CLINICAL TRIAL: NCT04277221
Title: Autologous Dendritic Cell / Tumor Antigen (ADCTA-SSI-G1) for Adjuvant Immunotherapy in Standard Treatment of Recurrent Glioblastoma Multiforme (GBM): A Multi-center, Open-label, Randomized Phase III Clinical Trial
Brief Title: ADCTA for Adjuvant Immunotherapy in Standard Treatment of Recurrent Glioblastoma Multiforme (GBM)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Safe Save Medical Cell Sciences & Technology Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADCTA-SSI-G1
Record Dates: First submitted 2020-02-14; First posted 2020-02-20 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Glioblastoma Multiforme
Keywords: Recurrent Glioblastoma Multiforme; Immunotherapy; Dendritic Cell
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard therapy with ADCTA vaccine (study group) (Experimental): - ADCTA vaccine as study treatment
  Dose(s): Ten doses, including 2~4×10^7 cells for the 1st dose (double doses), and 1~2×10^7cells for the 2nd to 10th doses.
  Administrative route: The ADCTA vaccine will be injected in axillar or inguinal regions close to lymphnodes subcutaneously at clinic.
  Frequency: The primary immunization inoculation is followed by 3 vaccines bi-weekly and then 6 vaccines monthly inoculation, for a total of 10 doses.
  - Bevacizumab as standard therapy
  Interventions: Biological: Autologous Dendritic Cell/Tumor Antigen, ADCTA
- Standard therapy (control group) (Active Comparator): * No study treatment
  * Bevacizumab as standard therapy
  Interventions: Biological: Autologous Dendritic Cell/Tumor Antigen, ADCTA

INTERVENTIONS:
Biological: Autologous Dendritic Cell/Tumor Antigen, ADCTA — ADCTA is an individualized cell immunotherapy co-culturing autologous dendritic cells derived from peripheral blood mononuclear cells (PBMNCs) with autologous tumor cell as antigen in order to evoke specific immune response.

SUMMARY:
To confirm the result of previous Phase I/II and phase II clinical trials, this trial is to test the efficacy and safety of ADCTA immunotherapy plus the standard therapy in comparison with standard therapy alone in patients with recurrent GBM.

ELIGIBILITY:
Inclusion Criteria:

1. Specimen collection screening

   * Karnofsky performance status (KPS) ≥ 60 at assessment prior to surgery
   * ≥ 18 and ≤ 70 years of age
   * Subject has been diagnosed with GBM and has undergone resection surgery followed by standard brain RT + concurrent temozolomide and adjuvant temozolomide, and progression occurred. The foregoing progression is defined as when patients with primary GBM experience an image or clinical deterioration after receiving standard of care.
   * Contrast-enhanced MRI suspects recurrent GBM
   * Supratentorial tumor
   * Must voluntarily sign and date informed consent form for specimen acquisition and future use, for study screening, approved by an Independent Ethics Committee (IEC)/ Institutional Review Board (IRB), prior to the initiation of any study-specific procedures
2. Study screening

   * Karnofsky performance status (KPS) ≥ 60 at randomization
   * Submission of fresh tumor
   * Post-operation contrast-enhanced MRI scan must be done after surgical resection, with the intent for cyto-reduction ≥ 80% of the contrast-enhancing tumor mass
   * Histologically confirmed WHO grade IV glioma by pathology tissue screening
   * Subjects receiving bevacizumab as standard of care for given indication
   * Subject has adequate bone marrow, renal, and hepatic function prior to randomization as follow:

     1. White blood cell (WBC) count ≥ 2,000/mm^3;
     2. Absolute neutrophil count (ANC) ≥ 1,000/mm^3;
     3. Platelets ≥ 100,000/mm^3;
     4. Hemoglobin (Hgb) ≥ 8.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dL is acceptable.);
     5. Blood Urea Nitrogen (BUN) < 30 mg/dL;
     6. Creatinine < 2 mg/dL;
     7. Renal function: calculated creatinine clearance ≥ 30 mL/min;
     8. Hepatic function: Total bilirubin ≤ 3 times upper limit of normal (ULN), Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2 times ULN;
     9. Prothrombin Time (PT) and activated partial thromboplastin time (PTT) ≤ 1.6 times ULN unless therapeutically warranted.
   * Subjects with recurrent GBM (Grade IV) are eligible for this protocol. An independent neuropathologist will review this diagnosis during the enrollment process
   * Must voluntarily sign and date informed consent form, for study participation, approved by an Independent Ethics Committee (IEC)/ Institutional Review Board (IRB), prior to the initiation of any study-specific procedures

Exclusion Criteria:

1. Specimen collection screening

   * Multifocal GBM
   * Prior invasive malignancy (except for non-melanomatous skin cancer; carcinoma in situ of breast, oral cavity or cervix) unless disease free for ≥ 2 years
   * Subject has used bevacizumab or immune checkpoint blockade to treat GBM
   * Lactating or pregnant female
   * Positive viral serology for HIV or syphilis at time of screening
2. Study screening

   * Subjects having a biopsy only at surgery or tumor cell insufficiency at preparation
   * Inability to undergo contrast-enhanced MRI scans
   * Subjects receiving investigational study drug for any indication or immunological-based treatment for any reason (Filgrastim may be used for prevention of severe neutropenia)
   * Inability to stop or decrease the use of corticosteroid doses to 4 mg/day prior to randomization
   * Tumor progression documented according to modified RANO criteria prior to randomization (approximately 5 weeks after surgery)
   * Severe, active comorbidity, defined as follow:

     1. Subject with clinically defined Acquired Immune-Deficiency Syndrome (AIDS)-defining illness;
     2. Subjects with acute hepatitis C or B infection;
     3. Severe hepatic impairment (Child-Pugh category C or higher);
     4. Electrocardiogram (ECG) with evidence of acute cardiac ischemia prior to randomization;
     5. Transmural myocardial infarction or ischemia prior to enrollment;
     6. Any other major medical illnesses or psychiatric impairments that in the Investigator's opinion will prevent administration or completion of protocol therapy
   * Subject used Gliadel wafer implant in surgery during screening process

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | The duration will be calculated from the date of randomization until the date of death from any cause, assessed up to 60 months.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | The duration will be calculated from the date of randomization until the date of first documented progression according to the modified RANO or date of death from any cause, whichever came first,assessed up to 60 months.
Progression-free Survival at 6 months (PFS6) | The duration will be calculated from the date of randomization to the date of the sixth month.
1 and 2-year Survival Rate | The duration will be calculated from the date of randomization to the date of the first year and the second year.

CONTACTS AND LOCATIONS:
Overall Officials: Peng-Wei Hsu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (7):
- Taiwan (7):
  - Chang Gung Memorial Hospital, Chiayi branch, Chiayi City
  - Chang Gung Memorial Hospital, Kaohsiung branch, Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung branch, Keelung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Chang Gung Memorial Hospital, Linkou branch, Taoyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chang CN, Huang YC, Yang DM, Kikuta K, Wei KJ, Kubota T, Yang WK. A phase I/II clinical trial investigating the adverse and therapeutic effects of a postoperative autologous dendritic cell tumor vaccine in patients with malignant glioma. J Clin Neurosci. 2011 Aug;18(8):1048-54. doi: 10.1016/j.jocn.2010.11.034. Epub 2011 Jun 28. PMID 21715171
- [Derived] Woroniecka K, Fecci PE. Immuno-synergy? Neoantigen vaccines and checkpoint blockade in glioblastoma. Neuro Oncol. 2020 Sep 29;22(9):1233-1234. doi: 10.1093/neuonc/noaa170. No abstract available. PMID 32691060